CLINICAL TRIAL: NCT05273541
Title: Beijing 302 Hospital
Brief Title: Safety and Immunogenicity of Prime-boost Vaccination of SARS-CoV-2 in Patients With Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ky-2021-7-9-2
Record Dates: First submitted 2022-02-23; First posted 2022-03-10 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-02

CONDITIONS: Patients With Cancer; Vaccine Reaction; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prime-boost vaccination (Experimental): Patients in the experimental group need to accept the prime-boost vaccination regimen
  Interventions: Biological: Coronavirus vaccination

INTERVENTIONS:
Biological: Coronavirus vaccination — Patients in this trial need to accept a prime-boost vaccination against SARS-CoV-2 after 6 to 8 months of the first vaccination

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection has caused a global pandemic since late 2019 that resulted in more than 360 million population infection. Patients with cancers may be at higher risk of infection and severity than those without cancer. Mass vaccination has been carried out, but reinfection and vaccine breakthrough cases still occur. Now, the prime-boost regimen was identified safe and efficient, but the reactogenicity and immunogenicity of prime-boost vaccine strategy in cancer patients were not known.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, open-label clinical trial. A total of 100 patients with different cancers including breast cancer, hepatocellular carcinoma, lung cancer, esophageal cancer, gastric cancer and colorectal cancer were included in this heterologous prime-boost vaccination study. All of the patients will further accept 12 months follow-up study after prime-boost vaccination. Safety, reactogenicity and immunogenicity of the prime-boost vaccination in those patients will be carefully recorded and detected.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years.
2. Patients with diagnosed cancers including breast cancer, hepatocellular carcinoma, lung cancer, esophageal cancer, gastric cancer and colorectal cancer.
3. Patients who have received local or systemic anti-cancer therapies according to the treatment guidelines previously or currently, and have a stable condition with the ECOG score below 2.
4. The functions of multi-organs were normal or basically normal, and there are no contraindications for vaccination.

Exclusion Criteria:

1. Patients with acute attack of chronic diseases.
2. Patients have history of convulsion, epilepsy, encephalopathy and psychosis. Patients who are allergic to any component of the vaccine, or have a serious history of vaccine allergy.
3. Pregnant or lactating women.
4. Sufferring serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, and severe hypertension can not be well controlled by drugs.

   Patients have severe chronic diseases or diseases can not be controlled well during the progress, such as asthma, diabetes, thyroid disease, etc. Congenital or acquired angioedema / neuroedema.
5. Systemic cytotoxic drugs, cell therapies including NK cells, cytokine induced killer cells, Dendritic cells, CTL and stem cells infusion are required during vaccination.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-11 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse effects after prime-boost vaccination | Within 1 week after the prime-boost vaccination
  Safety of the prime-boost vaccine
Titers of anti-SARS-CoV-2 antibodies | Within 3 months after the prime-boost vaccination
  Immunogenicity of prime-boost vaccine

SECONDARY OUTCOMES:
Occurence of adverse effects after prime-boost vaccination | Within 1 month after the prime-boost vaccination
  Safety of the prime-boost vaccine
Titers of anti-SARS-CoV-2 antibodies | Within 12 months after the prime-boost vaccination
  Immunogenicity of prime-boost vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Shu-juan Li, MD, Study Director — Beijing 302 Hospital
Locations (1):
- 302 Hospital, Beijing, China

REFERENCES:
- [Background] Lai CC, Wang JH, Hsueh PR. Population-based seroprevalence surveys of anti-SARS-CoV-2 antibody: An up-to-date review. Int J Infect Dis. 2020 Dec;101:314-322. doi: 10.1016/j.ijid.2020.10.011. Epub 2020 Oct 9. PMID 33045429
- [Background] Dai M, Liu D, Liu M, Zhou F, Li G, Chen Z, Zhang Z, You H, Wu M, Zheng Q, Xiong Y, Xiong H, Wang C, Chen C, Xiong F, Zhang Y, Peng Y, Ge S, Zhen B, Yu T, Wang L, Wang H, Liu Y, Chen Y, Mei J, Gao X, Li Z, Gan L, He C, Li Z, Shi Y, Qi Y, Yang J, Tenen DG, Chai L, Mucci LA, Santillana M, Cai H. Patients with Cancer Appear More Vulnerable to SARS-CoV-2: A Multicenter Study during the COVID-19 Outbreak. Cancer Discov. 2020 Jun;10(6):783-791. doi: 10.1158/2159-8290.CD-20-0422. Epub 2020 Apr 28. PMID 32345594
- [Background] Monin L, Laing AG, Munoz-Ruiz M, McKenzie DR, Del Molino Del Barrio I, Alaguthurai T, Domingo-Vila C, Hayday TS, Graham C, Seow J, Abdul-Jawad S, Kamdar S, Harvey-Jones E, Graham R, Cooper J, Khan M, Vidler J, Kakkassery H, Sinha S, Davis R, Dupont L, Francos Quijorna I, O'Brien-Gore C, Lee PL, Eum J, Conde Poole M, Joseph M, Davies D, Wu Y, Swampillai A, North BV, Montes A, Harries M, Rigg A, Spicer J, Malim MH, Fields P, Patten P, Di Rosa F, Papa S, Tree T, Doores KJ, Hayday AC, Irshad S. Safety and immunogenicity of one versus two doses of the COVID-19 vaccine BNT162b2 for patients with cancer: interim analysis of a prospective observational study. Lancet Oncol. 2021 Jun;22(6):765-778. doi: 10.1016/S1470-2045(21)00213-8. Epub 2021 Apr 27. PMID 33930323
- [Background] Fendler A, Au L, Shepherd STC, Byrne F, Cerrone M, Boos LA, Rzeniewicz K, Gordon W, Shum B, Gerard CL, Ward B, Xie W, Schmitt AM, Joharatnam-Hogan N, Cornish GH, Pule M, Mekkaoui L, Ng KW, Carlyle E, Edmonds K, Rosario LD, Sarker S, Lingard K, Mangwende M, Holt L, Ahmod H, Stone R, Gomes C, Flynn HR, Agua-Doce A, Hobson P, Caidan S, Howell M, Wu M, Goldstone R, Crawford M, Cubitt L, Patel H, Gavrielides M, Nye E, Snijders AP, MacRae JI, Nicod J, Gronthoud F, Shea RL, Messiou C, Cunningham D, Chau I, Starling N, Turner N, Welsh L, van As N, Jones RL, Droney J, Banerjee S, Tatham KC, Jhanji S, O'Brien M, Curtis O, Harrington K, Bhide S, Bazin J, Robinson A, Stephenson C, Slattery T, Khan Y, Tippu Z, Leslie I, Gennatas S, Okines A, Reid A, Young K, Furness AJS, Pickering L, Gandhi S, Gamblin S, Swanton C; Crick COVID-19 Consortium; Nicholson E, Kumar S, Yousaf N, Wilkinson KA, Swerdlow A, Harvey R, Kassiotis G, Larkin J, Wilkinson RJ, Turajlic S; CAPTURE consortium. Functional antibody and T cell immunity following SARS-CoV-2 infection, including by variants of concern, in patients with cancer: the CAPTURE study. Nat Cancer. 2021 Dec;2(12):1321-1337. doi: 10.1038/s43018-021-00275-9. Epub 2021 Oct 27. PMID 35121900
- [Background] Villarreal-Garza C, Vaca-Cartagena BF, Becerril-Gaitan A, Ferrigno AS, Mesa-Chavez F, Platas A, Platas A. Attitudes and Factors Associated With COVID-19 Vaccine Hesitancy Among Patients With Breast Cancer. JAMA Oncol. 2021 Aug 1;7(8):1242-1244. doi: 10.1001/jamaoncol.2021.1962. PMID 34110371
- [Background] Wang J, Hou Z, Liu J, Gu Y, Wu Y, Chen Z, Ji J, Diao S, Qiu Y, Zou S, Zhang A, Zhang N, Wang F, Li X, Wang Y, Liu X, Lv C, Chen S, Liu D, Ji X, Liu C, Ren T, Sun J, Zhao Z, Wu F, Li F, Wang R, Yan Y, Zhang S, Ge G, Shao J, Yang S, Liu C, Huang Y, Xu D, Li X, Ai J, He Q, Zheng MH, Zhang L, Xie Q, Rockey DC, Fallowfield JA, Zhang W, Qi X. Safety and immunogenicity of COVID-19 vaccination in patients with non-alcoholic fatty liver disease (CHESS2101): A multicenter study. J Hepatol. 2021 Aug;75(2):439-441. doi: 10.1016/j.jhep.2021.04.026. Epub 2021 Apr 24. PMID 33905793